CLINICAL TRIAL: NCT01314105
Title: Phase I Dose Escalation Trial to Determine the Maximum Tolerated Dose of BIBF 1120 in Combination With Carboplatin and Pegylated Liposomal Doxorubicin (PLD) in Patients With a First, Second or Third Platinum Sensitive Relapse of Advanced Epithelial Ovarian Cancer, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: BIBF 1120 + Carboplatin/Pegylated Liposomal Doxorubicin (PLD) in Patients With Advanced Ovarian Cancer, Fallopian Tube Carcinoma or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199.119; 2010-022523-30 (EudraCT Number)
Record Dates: First submitted 2011-03-08; First posted 2011-03-14 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Neoplasms; Peritoneal Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms | interventions — nintedanib; 1-dodecylpyridoxal

ARMS (3):
- BIBF 1120 L+ Carboplatin + PLD (Experimental): BIBF 1120 (100 mg twice daily (BID)) + Carboplatin (Area Under the Curve (AUC) 5 mg/mL*min) + PLD (30 mg/m2)
  Interventions: Drug: BIBF 1120 + PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min
- BIBF 1120 M + Carboplatin + PLD (Experimental): BIBF 1120 (150 mg twice daily (BID)) + Carboplatin (Area Under the Curve (AUC) 5 mg/mL*min) + PLD (30 mg/m2)
  Interventions: Drug: BIBF 1120 + PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min
- BIBF 1120 H + Carboplatin + PLD (Experimental): BIBF 1120 (200 mg twice daily (BID)) + Carboplatin (Area Under the Curve (AUC) 5 mg/mL*min) + PLD (30 mg/m2)
  Interventions: Drug: BIBF 1120+ PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min

INTERVENTIONS:
Drug: BIBF 1120 + PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min — BIBF1120 twice daily along with standard therapy of PLD + carboplatin
  Arms: BIBF 1120 M + Carboplatin + PLD
Drug: BIBF 1120+ PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min — BIBF1120 twice daily along with standard therapy of PLD + carboplatin
  Arms: BIBF 1120 H + Carboplatin + PLD
Drug: BIBF 1120 + PLD 30 mg/m2 + CBDCA AUC5 mg/mL*min — BIBF1120 twice daily along with standard therapy of PLD + carboplatin
  Arms: BIBF 1120 L+ Carboplatin + PLD

SUMMARY:
This phase I, open label dose escalation study will investigate the addition of BIBF 1120 to treatment with the combination of carboplatin and Pegylated Liposomal Doxorubicin (PLD) in patients with advanced, platinum sensitive relapsed ovarian cancer, fallopian tube carcinoma or primary peritoneal cancer.

ELIGIBILITY:
Inclusion criteria:

1. Female patients, age 18 years or older, with a first, second or third relapse of histologically (on initial diagnosis) confirmed epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal cancer
2. Up to three lines of prior chemo (chemotherapy before and after interval surgery to be counted as one line therapy), with treatment free interval of > 6 months (= time between last administration of prior anti-cancer treatment, including chemotherapy, hormonal therapy, or radiation therapy, and diagnosis of progressive disease)
3. Platinum based chemo in immediately preceding line
4. Eligibility for treatment with i.v. chemotherapy regimen of carboplatin AUC 5 and PLD 30 mg/m2 every 4 weeks
5. Life expectancy of at least 3 months
6. Written informed consent that is consistent with International Conference of Harmonisation (ICH)-Good Clinical Practice (GCP) guidelines
7. Eastern Cooperative Oncology Group (ECOG) performance score 0 or1
8. Prior treatment with angiogenesis inhibitor (bevacizumab, TKI inhibiting VEGFR-2) is allowed provided treatment with bevacizumab has been discontinued = 28 days prior to start of therapy and treatment with the TKI has been discontinued = 3 months prior to start of therapy, provided anti-angiogenic therapy was added to only one of the preceding lines of therapy

Exclusion criteria:

1. Prior chemotherapy with doxorubicin (any formulation, liposomal or non-liposomal doxorubicin).
2. Any contraindications for therapy with PLD or carboplatin, e.g. a history of hypersensitivity reactions to platinum-containing compounds and their excipients.
3. Hypersensitivity to active substance or to any of the excipients of BIBF 1120.
4. Treatment with other investigational drugs or participation in another clinical trial testing a drug within the past four weeks before start of therapy or concomitantly with this trial (exception: for previous treatment with angiogenesis inhibitors, cf. inclusion criterion #8).
5. Laboratory values indicating an increased risk for adverse events.
6. Major surgery within 4 weeks prior to start of study treatment.
7. Patients for whom surgery is planned, e.g. interval debulking surgery.
8. Clinically relevant non-healing wound, ulcer (intestinal tract, skin) or bone fracture.
9. Clinical symptoms or signs of gastrointestinal obstruction that require parenteral nutrition or hydration.
10. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug.
11. History of clinical symptoms of brain metastases.
12. Prior thrombosis or thromboembolic event in the presence of an inherited coagulopathy.
13. History of a cerebral vascular accident, transient ischemic attack or subarachnoid haemorrhage within the past 6 months.
14. Known inherited or acquired bleeding disorder.
15. Significant cardiovascular diseases.
16. Serious infections in particular if requiring systemic antibiotic (antimicrobial, antifungal) or antiviral therapy.
17. Other malignancy diagnosed within the past 5 years.
18. Known serious illness or concomitant non-oncological disease.
19. Patients unable to comply with the protocol.
20. Patients with preserved reproductive capacity who are sexually active and unwilling to use a medically acceptable method of contraception.
21. Pregnancy or breast feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03-15 (Actual); Primary Completion 2013-07-29 (Actual); Study Completion 2016-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Abbreviations Used:
  CTCAE: Common Terminology Criteria for Adverse Events
  ALT: Alanine Amino Transferase
  AST: Aspartate Aminotransferase
  ULN: Upper Limit of Normal
Groups:
- Nintedanib 150mg: Nintedanib (150 mg twice daily (BID), except the day of chemotherapy infusion) administered orally plus standard therapy of carboplatin (Area Under the Curve (AUC) 5 mg/mL*min) and PLD (30 mg/m2) which were administered by intravenous infusion once every 28 days.
- Nintedanib 200mg: Nintedanib (200 mg twice daily (BID), except the day of chemotherapy infusion) administered orally plus standard therapy of carboplatin (Area Under the Curve (AUC) 5 mg/mL*min) and PLD (30 mg/m2) which were administered by intravenous infusion once every 28 days.
Period: Overall Study
Arm/Group | Nintedanib 150mg | Nintedanib 200mg
Started | 7 | 12
Completed | 0 | 0
Not Completed | 7 | 12
Not completed — Progressive Disease | 6 | 10
Not completed — Refused to continue taking medication | 0 | 1
Not completed — Other Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS) which included all patients who were administered at least one dose of any study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib 150mg | Nintedanib 200mg | Total
Number analyzed (Participants) | 7 | 12 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (12.7) [36 to 71] | 53.1 (6.4) [40 to 63] | 54.9 (9.2) [36 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Nintedanib Based on the Occurrence of DLTs During Treatment Course 1
Description: Maximum Tolerated Dose (MTD) of nintedanib in combination with carboplatin and pegylated liposomal doxorubicin based on the occurrence of dose limiting toxicities (DLTs) during treatment course 1. MTD will be determined among the first 6 evaluable patients in each dose level. MTD is the highest dose at which the incidence of DLT is less than 2/6.
Time Frame: First 28-day treatment cycle
Population: MTD set which included patients in the dose escalation part of the trial who started treatment course 2 and/or took 1 dose of carboplatin and PLD, started nintedanib (nin) and did not miss more than 13 doses of nin and/or took 1 dose of carboplatin and PLD, started nin and discontinued treatment due to a dose limiting toxicity during the MTD period
Measure: Number; unit: mg
Arm/Group | Nintedanib 150mg | Nintedanib 200mg
Number analyzed (Participants) | 6 | 6
mg | NA — MTD was not determined for this dose group | 200

2. Primary Outcome: Dose Limiting Toxicities During Treatment Course 1
Description: Number of patients with dose limiting toxicity (DLT) occurring during treatment course 1
  The following AEs were to be reported as DLT events if their occurrence was considered to be drug-related:
  Haematological toxicity:
  * Any CTCAE grade 4 haematological toxicity
  * CTCAE grade 4 neutropenia that was not associated with fever ≥38.5°C, if persisting for >7 days despite adequate supportive treatment
  * CTCAE grade ≥3 neutropenia of any duration if associated with fever ≥38.5°C
  * Any CTCAE grade 4 thrombocytopenia
  * CTCAE grade ≥3 thrombocytopenia if associated with bleeding of CTCAE grade ≥2
  Non-haematological toxicity:
  * CTCAE grade ≥3 diarrhoea despite optimal medical management
  * CTCAE grade 2 diarrhoea persisting for more than 7 days despite optimal medical management
  * CTCAE grade ≥2 vomiting despite optimal medical management
  * ALT and/or AST elevation of CTCAE grade ≥3
  * ALT and/or AST elevation of >3x ULN in conjunction with bilirubin increase >2x ULN
Time Frame: First 28-day treatment cycle
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nintedanib 150mg | Nintedanib 200mg
Number analyzed (Participants) | 6 | 6
participants | 1 | 1

3. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Nintedanib
Description: Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-inf) of nintedanib during course 1 and course 2
Time Frame: 5 minutes (min) before drug administration and 1 hour (h) 2h, 3h, 4h, 6h, 8h, 10h, 24h, 144h, 312h and 456h after drug administration
Population: Pharmacokinetic (PK) set: All patients in the treated set who were documented to have received at least one dose of nintedanib and who had at least one valid pharmacokinetic parameter concentration available
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/millilitre (ng*h/mL)
Arm/Group | Nintedanib 150mg | Nintedanib 200mg
Number analyzed (Participants) | 7 | 12
nanogram*hour/millilitre (ng*h/mL)
  Treatment Course 1 (150mg: N=5; 200mg: N=10) | 335 (88.5) | 482 (38.8)
  Treatment Course 2 (150mg: N=7) | 482 (76.1) | NA (NA) — Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Drug Concentration (AUC0-tz) of Nintedanib
Description: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable drug concentration (AUC0-tz) of nintedanib during course 1 and course 2.
Time Frame: as for outcome 3
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib 150mg | Nintedanib 200mg
Number analyzed (Participants) | 7 | 12
ng*h/mL
  Treatment Course 1 (150mg: N=6; 200mg: N=11) | 283 (70.2) | 422 (36.9)
  Treatment Course 2 (150mg: N=8; 200mg: N=7) | 406 (59.0) | 476 (37.6)

5. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) of Nintedanib
Description: Maximum measured plasma concentration (Cmax) of nintedanib during course 1 and course 2
Time Frame: as for outcome 3
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib 150mg | Nintedanib 200mg
Number analyzed (Participants) | 7 | 12
ng/mL
  Treatment Course 1 (150mg: N=6; 200mg: N=11) | 38.8 (40.3) | 69.0 (27.9)
  Treatment Course 2 (150mg: N=8; 200mg: N=7) | 65.8 (51.6) | 82.2 (43.0)

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Carboplatin (Determined as Total Platinum)
Description: Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-inf) of carboplatin (determined as total platinum) during treatment course 1 and course 2.
Time Frame: 5 minutes (min) before drug administration and 30 min,59 min, 1 hour (h) 15 min, 1h 29min, 1h 45min, 2h 15min, 2h 45min, 4h, 6h, 7h 30min, 9h, 23h 55min, 26h, 28h, 32h, 48h, 168h, 336h and 480h after drug administration
Population: PK set.Goal is to find MTD for nintedanib,two doses of nintedanib separately displayed.However carboplatin,PLD are given as background,therefore only measured to know exposure.As result displaying all subjects is sufficient.Further we decided to make separate table for MTD dose(200mg nintedanib).Separate table for 150mg nintedanib doesnt add value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- All Patients: Nintedanib (200 mg or 150 mg twice daily (BID), except the day of chemotherapy infusion) administered orally plus standard therapy of carboplatin (Area Under the Curve (AUC) 5 mg/mL*min) and PLD (30 mg/m2) which were administered by intravenous infusion once every 28 days.
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 12 | 19
ng/mL
  Treatment Course 1 (200mg:N=10; All Patients:N=16) | 271000 (15.1) | 267000 (15.1)
  Treatment Course 2 (200mg:N=7; All Patients:N=16) | 325000 (15.4) | 324000 (14.7)

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero Extrapolated to Infinity (AUC 0-inf) of Carboplatin During Treatment Course 1 and Course 2 (Determined as Ultrafilterable Platinum)
Description: Area under the plasma concentration-time curve over the time interval from zero extrapolated to infinity (AUC 0-inf) of carboplatin during treatment course 1 and course 2 (determined as ultrafilterable platinum).
  Geometric mean (gMean) and Geometric coefficient of Variation (gCV) were not calculable for treatment course 2 as 2/3 of patients had quantifiable values.
Time Frame: 5 minutes (min) before drug administration and 30 min,59 min, 1 hour (h) 15 min, 1h 29min, 1h 45min, 2h 15min, 2h 45min, 4h, 6h, 7h 30min, 9h, 23h 55min, 25h, 26h, 27h, 28h, 30h, 32h, and 34h after drug administration
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 9 | 19
ng*h/mL
  Treatment Course 1 (200mg:N=9; All Patients:N=16) | 71000 (69.3) | 70700 (107)
  Treatment Course 2 (200mg:N=NA; All Patients:N=NA) | NA (NA) — Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | NA (NA) — Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules.

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Drug Concentration (AUC0-tz) of Carboplatin (Determined as Total Platinum)
Description: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable drug concentration (AUC0-tz) of carboplatin during course 1 and course 2 (determined as total platinum).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 12 | 19
ng*h/mL
  Treatment Course 1 (200mg:N=10; All Patients:N=16) | 223000 (18.4) | 220000 (17.1)
  Treatment Course 2 (200mg:N=7; All Patients:N=16) | 258000 (15.8) | 260000 (14.7)

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Drug Concentration (AUC0-tz) of Carboplatin (Determined as Ultrafilterable Platinum)
Description: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable drug concentration (AUC0-tz) of carboplatin during course 1 and course 2 (determined as ultrafilterable platinum).
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 12 | 19
ng*h/mL
  Treatment Course 1 (200mg:N=9; All Patients:N=16) | 58500 (26.0) | 53800 (26.7)
  Treatment Course 2 (200mg:N=6; All Patients:N=15) | 56200 (26.5) | 55700 (29.8)

10. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) of Carboplatin (Total Platinum)
Description: Maximum measured plasma concentration (Cmax) of carboplatin during course 1 and course 2 (determined as total platinum).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 12 | 19
ng/mL
  Treatment Course 1 (200mg:N=10; All Patients:N=16) | 24600 (49.1) | 24000 (37.7)
  Treatment Course 2 (200mg:N=7; All Patients:N=16) | 27100 (22.7) | 23900 (25.2)

11. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) of Carboplatin During Course 1 and Course 2 (Determined as Ultrafilterable Platinum)
Description: Maximum measured plasma concentration (Cmax) of carboplatin during course 1 and course 2 (determined as ultrafilterable platinum).
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 12 | 19
ng/mL
  Treatment Course 1 (200mg:N=9; All Patients:N=16) | 26000 (48.4) | 24600 (38.0)
  Treatment Course 2 (200mg:N=6; All Patients:N=15) | 27000 (26.6) | 24400 (23.0)

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero Extrapolated to Infinity (AUC 0-inf) of PLD (Determined as Total Plasma Doxorubicin) During Treatment Course 1 and Course 2
Description: Area under the plasma concentration-time curve over the time interval from zero extrapolated to infinity (AUC 0-inf) of pegylated liposomal doxorubicin (PLD) (determined as total plasma doxorubicin) during treatment course 1 and course 2.
  Geometric mean (gMean) and Geometric coefficient of Variation (gCV) were not calculable for treatment course 1 as for only 2 patients evaluable concentrations were available.
Time Frame: 5 minutes (min) before drug administration and 30 min,59 min, 1 hour (h) 15 min, 1h 29min, 1h 45min, 2h 15min, 2h 45min, 4h, 6h, 7h 30min, 9h, 25h, 27h, 30h, 34h, 48h, 168h, 336h and 480h after drug administration
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 3 | 19
µg*h/mL
  Treatment Course 1 (200mg:N=NA; All Patients:N=8) | NA (NA) — Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | 2280 (20.1)
  Treatment Course 2 (200mg:N=3; All Patients:N=10) | 2120 (38.4) | 2300 (25.5)

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Drug Concentration (AUC0-tz) of PLD (Determined as Total Plasma Doxorubicin) During Treatment Course 1 and Course 2
Description: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable drug concentration (AUC0-tz) of pegylated liposomal doxorubicin (PLD) (determined as total plasma doxorubicin) during treatment course 1 and course 2.
  Geometric mean (gMean) and Geometric coefficient of Variation (gCV) were not calculable for treatment course 1 as for only 2 patients evaluable concentrations were available.
Time Frame: as for outcome 12
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 3 | 19
µg*h/mL
  Treatment Course 1 (200mg:N=NA; All Patients:N=8) | NA (NA) — Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | 2230 (19.3)
  Treatment Course 2 (200mg:N=3; All Patients:N=10) | 2060 (35.2) | 2210 (24.8)

14. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) of PLD (Determined as Total Plasma Doxorubicin) During Treatment Course 1 and Course 2
Description: The maximum measured plasma concentration (Cmax) of pegylated liposomal doxorubicin (PLD) (determined as total plasma doxorubicin) during treatment course 1 and course 2.
  Geometric mean (gMean) and Geometric coefficient of Variation (gCV) were not calculable for treatment course 1 as for only 2 patients evaluable concentrations were available.
Time Frame: as for outcome 12
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 3 | 19
µg/mL
  Treatment Course 1 (200mg:N=NA; All Patients:N=8) | NA (NA) — Not calculated as reliable estimation can only be performed when at least 2/3 of the data are available and thus the gMean and gCV is not calculated according to internal rules. | 18.9 (14.5)
  Treatment Course 2 (200mg:N=3; All Patients:N=8) | 19.0 (13.5) | 19.0 (18.0)

15. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero Extrapolated to Infinity (AUC 0-inf) of PLD (Determined as Plasma Doxorubicinol)
Description: Area under the plasma concentration-time curve over the time interval from zero extrapolated to infinity (AUC 0-inf) of pegylated liposomal doxorubicin (PLD) (determined as plasma doxorubicinol).
  Due to interference from doxorubicin, doxorubicinol concentrations could not be determined and doxorubicinol PK parameters could not be evaluated.
Time Frame: as for outcome 12
Population: as for outcome 6
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Drug Concentration (AUC0-tz) of PLD (Determined as Plasma Doxorubicinol)
Description: Area under the plasma concentration-time curve from time zero to the time of the last quantifiable drug concentration (AUC0-tz) of pegylated liposomal doxorubicin (PLD) (determined as plasma doxorubicinol).
  Due to interference from doxorubicin, doxorubicinol concentrations could not be determined and doxorubicinol PK parameters could not be evaluated.
Time Frame: as for outcome 12
Population: as for outcome 6
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) of PLD (Determined as Plasma Doxorubicinol)
Description: The maximum measured plasma concentration (Cmax) of pegylated liposomal doxorubicin (PLD) (determined as plasma doxorubicinol).
  Due to interference from doxorubicin, doxorubicinol concentrations could not be determined and doxorubicinol PK parameters could not be evaluated.
Time Frame: as for outcome 12
Population: as for outcome 6
Arm/Group | Nintedanib 200mg | All Patients
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Incidence and Intensity of Adverse Events
Description: Safety of nintedanib as indicated by intensity and incidence of adverse events, graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0.
  The CTCAE grades are the worst grade per patient. The CTCAE grades are Grade 1 as mild AE, Grade 2 as moderate AE, Grade 3 as severe AE, Grade 4 as lifethreatening or disabling AE, and Grade 5 as death related to AE.
Time Frame: From the first drug administration until 28 days after the last drug administration, up to 31 months
Population: Treated Set
Measure: Number; unit: participants
Arm/Group | Nintedanib 150mg | Nintedanib 200mg
Number analyzed (Participants) | 7 | 12
participants
  Grade 1 | 0 | 0
  Grade 2 | 2 | 0
  Grade 3 | 3 | 9
  Grade 4 | 2 | 3
  Grade 5 | 0 | 0

19. Secondary Outcome: Change From Baseline in Safety Laboratory Parameters
Description: Change from baseline in safety laboratory parameters.
Time Frame: From the first drug administration until 28 days after the last drug administration, up to 31 months
Population: Treated Set
Measure: Number; unit: percentage of participants
Arm/Group | Nintedanib 150mg | Nintedanib 200mg
Number analyzed (Participants) | 7 | 12
percentage of participants
  Alanine aminotransferase increased | 57.1 | 91.7
  Aspartate aminotransferase increased | 71.4 | 91.7
  Gamma-glutamyltransferase increased | 42.9 | 66.7
  Platelet count decreased | 28.6 | 58.3
  Blood alkaline phosphatase | 28.6 | 0
  Blood lactate dehydrogenase increased | 28.6 | 16.7
  Blood alkaline phosphatase increased | 14.3 | 25.0
  Haemoglobin decreased | 0 | 16.7
  Neutrophil count decreased | 0 | 16.7
  Blood bilirubin increased | 14.3 | 8.3
  Blood creatinine decreased | 14.3 | 0
  Gamma-glutamyltransferase | 14.3 | 0
  Haemoglobin | 14.3 | 0
  Neutrophil count | 14.3 | 0
  White blood cell count decreased | 14.3 | 0
  Amylase increased | 0 | 8.3
  Blood creatinine increased | 0 | 8.3
  Platelet count increased | 0 | 8.3

ADVERSE EVENTS:
Time Frame: From the first drug administration until 28 days after the last drug administration, up to 31months
Arm/Group | Nintedanib 150mg | Nintedanib 200mg
Serious Adverse Events (participants affected / at risk) | 3/7 | 4/12
Other Adverse Events (participants affected / at risk) | 6/7 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 150mg (N=7) | Nintedanib 200mg (N=12)
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib 150mg (N=7) | Nintedanib 200mg (N=12)
Anaemia (Blood and lymphatic system disorders) | 5 | 9
Leukopenia (Blood and lymphatic system disorders) | 5 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Xerophthalmia (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 11
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 12
Odynophagia (Gastrointestinal disorders) | 0 | 3
Oral pain (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 3
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 11
Asthenia (General disorders) | 6 | 11
Catheter site erythema (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Mucosal dryness (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 3 | 7
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 6
Xerosis (General disorders) | 1 | 0
Deficiency of bile secretion (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Allergy to animal (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Angular cheilitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 4
Parotitis (Infections and infestations) | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 11
Amylase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 11
Blood alkaline phosphatase (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 3
Blood bilirubin increased (Investigations) | 1 | 1
Blood creatinine decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 2
Gamma-glutamyltransferase (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 8
Haemoglobin (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 2
Neutrophil count (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 2 | 7
Platelet count increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3
Dysgeusia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 5 | 5
Paraesthesia (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 3
Choluria (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to interference from doxorubicin, doxorubicinol concentrations could not be determined and doxorubicinol PK parameters could not be evaluated.

Statistics of PK parameters are only estimated when at least 2/3 of the data are evaluable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.